CLINICAL TRIAL: NCT06053463
Title: Evaluation of Soft Multifocal Lenses in Presbyopic Previous Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Fogt (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Fogt, Principal Investigator, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023H0245
Record Dates: First submitted 2023-09-12; First posted 2023-09-25 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Presbyopia
Keywords: contact lenses; Multifocal contact lenses
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lens wear experience (Experimental): Subject will wear contact lenses for about a month during the day.
  Interventions: Device: Daily disposable multifocal soft contact lens

INTERVENTIONS:
Device: Daily disposable multifocal soft contact lens — Daily disposable multifocal soft contact lens that will be worn for 1 month.

SUMMARY:
To explore the wear experience in Dailies TOTAL1 Multifocal contact lenses in presbyopic adults who have previously dropped out of contact lens wear.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the wear experience of people with presbyopia who previously dropped out of contact lens wear when fit with a Delefilcon A soft lens multifocal lens. Investigators expect to enroll a relatively equal amount of former soft multifocal contact lens wearers who dropped out due to poor vision at distance or near and single vision wearers who dropped out due to poor near vision. The key endpoints include Visual Analog Scale survey of lens wear symptoms (comfort, dryness, vision) with contact lenses and assessment of the participant's quality of life with the Dailies TOTAL1 Multifocal® contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent.
* Any gender.
* Any racial or ethnic origin.
* At least 38 years of age or older.
* Willing to spend time for the study. Three visits are required to complete the study, and additional follow up visits could be scheduled if needed.
* Subjects must have corrected distance visual acuity in both eyes equivalent to 20/25 or better at the screening visit.
* Spectacle sphere power range between +6.00 to -10.00.
* Previously dropped out of contact lens wear due to vision or vision and discomfort.
* Good general health (defined by medication use that has not changed within the last month and the absence of medical conditions or treatments that are deemed confounding to the data as determined by the PI

Exclusion Criteria:

* Current or active ocular inflammation or infection as determined by the Investigator.
* Astigmatism ≥ 1.00 D in either eye.
* History of previous eye surgery.
* Strabismus or binocular vision abnormalities that prevent completion of testing, at the discretion of the Investigator.
* Demonstration or history of corneal ectasia or keratoconus.
* Pregnant or lactating

Min Age: 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Fogt, OD, MS, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - The Ohio State University College of Optometry, Columbus, Ohio
  - ProCare Vision Center, Granville, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lens Wear Experience
Started | 35
Completed | 25
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Lens Wear Experience
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale
Description: Visual Analog Scale survey of lens wear symptoms (vision) with contact lenses; percentage of participants with positive scores (> 50).
Time Frame: 1 month
Population: Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Lens Wear Experience
Number analyzed (Participants) | 25
Participants | 22

2. Primary Outcome: Quality of Life Survey
Description: Assessment of the participant's quality of life with the daily disposable multifocal contact lenses; percentage of participants with VAS scores greater than 50 on satisfaction survey.
Time Frame: 1 month
Population: Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Lens Wear Experience
Number analyzed (Participants) | 24
Participants | 22

ADVERSE EVENTS:
Time Frame: During the entirety of study participation. About 1 month.
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Lens Wear Experience
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT06053463/Prot_SAP_001.pdf